CLINICAL TRIAL: NCT03494205
Title: Urtica Comp. Gel for Prevention and Therapy of Radiation Dermatitis (An Interdisciplinary, Interprofessional Phase II Randomized Controlled Trial in Patients With Breast Cancer)
Brief Title: Urtica Comp. Gel for Prevention and Therapy of Radiation Dermatitis
Acronym: Urticacomp
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 211820931
Record Dates: First submitted 2018-02-22; First posted 2018-04-11 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Radiation Dermatitis
Keywords: Radiation Dermatitis; Urtica comp.
MeSH Terms: conditions — Radiodermatitis

STUDY DESIGN:
Intervention Model Description: randomized parallel design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test group (Experimental): For the patients of the test-group Urtica comp gel is applied three times per day locally on the skin as soon as the patient senses "itching, tingling" and/or reddening. Otherwise the skincare is exactly as the control group in line with the departments general guidelines.
  In case of marked worsening, e.g. epitheliolysis, the patient may receive "Flammazine and Ialugen plus" as rescue-care.
  Rescue care: according to the departments therapeutic guidelines patients will receive "Flammazine and/or Ialugen plus" as clinically indicated at the discretion of the treating physician (usually in cases of marked worsening of the skin condition like e.g. epitheliolysis).
  Interventions: Drug: Urtica comp. gel
- Control group (Active Comparator): Control group receiving the institutional standard skin care "Excipial-Hydrolotion" - all other therapeutic interventions, assessments and rescue-care will be the same in both groups.
  Interventions: Drug: institutional standard skin care "Excipial-Hydrolotion"

INTERVENTIONS:
Drug: Urtica comp. gel — Urtica comp. gel is a Swissmedic registered medication. The scope of application of Urtica comp. is an imbalanced, affected process of skin-regeneration, in particular when stemming from an overdose of heat or light.
  It is applied in first and second-degree burn and scalding, sunburn, allergic and hyperergic (excessive) skin conditions (dermatoses), insect bites, abrasions and ulcers.
  Other Names: Wund- und Brand Gel
  Arms: Test group
Drug: institutional standard skin care "Excipial-Hydrolotion" — The institutional standard skin care "Excipial-Hydrolotion" is available to all patients
  Other Names: Excipial
  Arms: Control group

SUMMARY:
A randomized controlled trial comparing Urtica comp. gel (Swissmedic listed medication in the category of "Anthroposophic Medication without Indication") against standard skin care, examining its effect in prevention and treatment of radiation dermatitis in breast cancer patients under Radiation therapy.

DETAILED DESCRIPTION:
Radiation dermatitis is one of the most common side effects of radiotherapy for cancer and affects around 95 % of patients receiving radiotherapy. Patients with breast cancer as well as patients with head and neck cancer are most frequently affected, due to the higher radiation dose to the skin, as compared to other cancer types.

Radiation dermatitis has a profound impact on the quality of a patient's life, due to pain and discomfort. Skin lesions bear a marked risk of infection. In addition, all these issues may be the cause of interruption of radiation therapy, resulting in inadequate disease treatment.

Despite a plentitude of studies researching local and systemic therapeutic approaches, currently no treatment (aside from local steroids which bear substantial side-effects) can be explicitly recommended.

Thus, further research, especially in therapeutic options with a positive side-effect spectrum would be highly beneficial.

Urtica comp. gel is a Swissmedic registered medication. It is e.g. applied in first and second-degree burn and scalding as well as sunburn and has been used in over 80 years with an excellent safety profile. Positive clinical experience in treating radiation dermatitis with Urtica comp. gel suggest studying this therapeutic option in a pilot trial.

ELIGIBILITY:
Inclusion Criteria:

* Radiation therapy for Breast Cancer
* Age >= 18 years
* Written informed consent

Exclusion Criteria:

* Ulcerated cancer at beginning of radiation therapy
* Skin lesions in the radiation area before start of radiation therapy
* Known allergies, hypersensitivity or reactions against one of the constituents of the investigational product [5]
* Any neurological or psychiatric conditions that, in the evaluation of the treating physician, deem the patient incapable to participate in the study
* Other clinically significant concomitant disease states (e.g., renal failure, hepatic dysfunction, cardiovascular disease, etc.) as judged by the PI

The following criteria are exclusion criteria for the conduct of the radiation therapy, which is prerequisite for inclusion into the study. Thus, such patients will anyway not meet the inclusion criteria and are explicitly excluded from participation:

* Women who are pregnant or breast feeding
* Lack of safe contraception, defined as: Female participants of childbearing potential, not using and not willing to continue using a medically reliable method of contraception for the entire study duration, such as oral, injectable, or implantable contraceptives, or intrauterine contraceptive devices, or who are not using any other method considered sufficiently reliable by the investigator in individual cases.
* Please note that female participants who are surgically sterilised / hysterectomised or post-menopausal for longer than 2 years are not considered as being of child bearing potential.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-05-02 (Actual); Primary Completion 2022-02-10 (Actual); Study Completion 2022-02-10 (Actual)

PRIMARY OUTCOMES:
Incidence of Radiation Dermatitis (RD) measured by the CTCAE | During the whole study (six weeks of therapy plus follow-up of six weeks)
  Comparison between both arms
Severity of RD measured by the CTCAE | During the whole study (six weeks of therapy plus follow-up of six weeks)
  Comparison between both arms

SECONDARY OUTCOMES:
Percentage of patients requiring no additional therapy for RD (e.g. Flammazine or Ialugen plus) | During the whole study (six weeks of therapy plus follow-up of six weeks)
  Comparison between both arms measuring the use of Flammazine or Ialugen plus (rescue-care)
Percentage of patients RD free at end of therapy (EOT) measured by the CTCAE | EOT (=time point specifically at end of 6 weeks of radiation therapy)
  Comparison between both arms
Percentage of patients with secondary skin infection / need of topical and systemic antibiotics | During the whole study (six weeks of therapy plus follow-up of six weeks)
  Comparison between both arms
Patients quality of life measured by the Skindex | During the whole study (six weeks of therapy plus follow-up of six weeks)
  Comparison between both arms.
Patients evaluation of the treatment (satisfaction) measured by the FACIT-TS-G (total scale) | EOT (=time point specifically at end of 6 weeks of radiation therapy)
  Comparison between both arms. The FACIT-TS-G (Functional Assessment of Chronic Illness Therapy treatment satisfaction - General) assesses the patients treatment satisfaction at the end of therapy (EOT after 6 weeks of Radiation therapy).
  The questionnaire consists of 8 questions, 3 of which are answered on a scale ranging from 0 (much worse) to 4 (much better), 3 questions ranging from 0 (not al all) to 3 (totally) and two questions which can be answered with 0 (no), 1(maybe) and 2 (yes). Thus on all scales a higher value represents a better outcome. The total score range is 0 (not satisfied at all) to 25 (highly satisfied).
Patients evaluation of the treatment (Skin condition) measured by visual analog scale (VAS) | During the whole study (six weeks of therapy plus follow-up of six weeks)
  with the Skin Condition VAS the patient self-assesses the skin condition in the radiation area.
  The questionnaire consists of 5 subscales: pain, itching, burning, irritation, visual appearance. Each scale ranges from 0 (not apparent) to 100 (worst possible expression). For the total score all values are summed up and divided by 5 (number of scales) resulting in a total score ranging from 0 (best possible outcome = no skin affection due to radiation) to 100 (worst possible outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Ursula Wolf, Study Director — University Bern, Institution of Complementary Medicine; Nikola Cihoric, MD PhD, Principal Investigator — University Bern, Department of Radiation Oncology
Locations (1):
- Universitätsklinik für Radio-Onkologie, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No
Individual Patient data will not be shared.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-01): https://cdn.clinicaltrials.gov/large-docs/05/NCT03494205/Prot_SAP_000.pdf